CLINICAL TRIAL: NCT05119010
Title: A Pilot Study Evaluating a Ketogenic Diet Concomitant to Nivolumab and Ipilimumab in Patients With Metastatic Renal Cell Carcinoma
Acronym: KETOREIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges: competition with another microbiome trial, patient refusal to join a dietary intervention study, poor tolerance of oral DPD (Grade 2 mucositis), and issues with organizing biological sample collection.
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A03550-39; 2020/3206 (Other: CSET number)
Record Dates: First submitted 2021-10-21; First posted 2021-11-12 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — 3-Hydroxybutyric Acid; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Patients will be included sequentially in each arm from arm A to arm D. When the first inclusion arm A will be full with 15 patients who passed the screening, then next patients will be enrolled in arm B, then it will be the same process with arm C and last patients will be included in arm D.
  However, the clinician has the option of including the patient in the standard diet arms with or without BHB (arm C or D), instead of the ketogenic diet arms (arm A or B), if the patient's organizational constraints do not allow for a strict ketogenic diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (Experimental): patients will be asked to follow in a continuous way a very low-carbohydrate, high-fat diets, which strictly limit carbohydrate consumption (less than 40g / day) and allow unlimited consumption of high-fat foods, such as pork belly, butter, coconuts oils, fat meat, eggs and cheese, etc… (cf appendix A). Patients will be provided with 2 meals (lunch and dinner), every meal with 2 dishes (first course and main course) and bread for every day for 3 months (ELIOR partnership).
  Interventions: Dietary Supplement: Continuous ketogenic diet
- B (Experimental): patients will be asked to follow in a discontinuous way (15 days on, 15 days off) a very low-carbohydrate, high-fat diets, which strictly limit carbohydrate consumption (less than 40g / day) and allow unlimited consumption of high-fat foods, such as pork belly, butter, coconuts oils, fat meat, eggs and cheese…etc (cf appendix A). Patients will be provided with 2 meals (lunch and dinner), every meal with 2 dishes (first course and main course) and bread for every day for the ketogenic diet period for 3 months (ELIOR partnership).
  Interventions: Dietary Supplement: Discontinuous ketogenic diet
- C (Experimental): patients will receive oral liquid ketone supplement BHB monoester, 2 tablespoons three times per day (depending on patient weight: at least 1g/kg weight body/day) 15 days-on 15 days off during 3 months. We would recommend taking it at least 30 to 60 min before meal times and they will receive standard diet (without any diet restrictions).
  Interventions: Dietary Supplement: beta-hydroxybutyrate (BHB) supplementation
- D (No Intervention): patients will receive standard diet (without any diet restrictions) and be followed up as in arms A, B, C.

INTERVENTIONS:
Dietary Supplement: Continuous ketogenic diet — ARM A : continuous ketogenic diet
  Arms: A
Dietary Supplement: Discontinuous ketogenic diet — ARM B : discontinuous ketogenic diet
  Arms: B
Dietary Supplement: beta-hydroxybutyrate (BHB) supplementation — ARM C : BHB supplementation
  Arms: C

SUMMARY:
The purpose of this study is to assess objective response rate (partial and complete response) of Nivolumab and Ipilimumab concomitant to a special diet (ketogenic diet, continuous or discontinuous) or standard diet with or without BHB according to RECIST v1.1 at 8 weeks.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving informed consent will undergo a 10 days screening period to determine eligibility for study entry. At week1day1, patients who meet the eligibility requirements will be enrolled in to :

* Arm A : continuous ketogenic diet for 3 months
* Arm B : discontinuous ketogenic diet (15 days on, 15 days off) for 3 months
* Arm C : oral liquid ketone supplement BHB monoester, 15 days-on 15 days off during 3 months.
* Arm D : standard diet (without any diet restrictions). and follow up as in arms A, B, C.

All patients will receive Nivolumab plus Ipilimumab according to practical routine.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women ≥ 18 years
2. Patients with a histologically confirmed Renal Cell Carcinoma with a clear-cell component, sarcomatoid or rhabdoid
3. Patients with metastatic (AJCC stage IV) Renal Cell Carcinoma, with at least one measurable lesion by CT Scan or MRI according to RECIST 1.1 or with clinically apparent disease that can be reliably monitored by the investigator
4. Patients who have not received a prior systemic therapy. Prior cytokine therapies (e.g. interleukine-2, interferon-α), vaccine therapy are allowed.
5. Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
6. Intermediate or poor risk group patients measured by the IMDC model
7. Patients with brain metastases will be eligible if they are: asymptomatic, without edema, not on corticosteroids more than 10 mg per day or already treated
8. Patients treated with radiation therapy will be eligible if they are: palliative, on focal radiation therapy, on immunosuppressive doses of systemic corticosteroids less than 10 mg per day.
9. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed
10. Patient should be able and willing to comply with study visits and procedures as per protocol
11. Patients must be affiliated to a social security system or beneficiary of the same
12. Women of childbearing potential must have a negative serum pregnancy test done within 24 hours prior to diet initiation. Potentially reproductive patients must agree to use an effective contraceptive method or practice adequate methods of birth control or practice complete abstinence while on treatment with Nivolumab and Ipilimumab
13. Women who are breastfeeding should discontinue nursing prior to the first dose of study drug and until 6 months after the last dose

Exclusion Criteria:

1. Weight loss > 5% in the last month
2. Weight loss > 10% during last 6 months
3. Albumin <30 g/l
4. Known or underlying medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would make the administration of study drug hazardous to the patient or obscure the interpretation of toxicity determination or adverse events.
5. Fatty acid oxidation disturbances
6. Uncontrolled diabetes defined as a hemoglobin A1C level > 8%. Diabetes is not exclusionary provided the patient is not maintained with either oral medications or insulin.
7. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements as determined by study team members.
8. Failure to submit to study clinical and biological follow-up for medical, geographic or social reasons
9. Pregnant or breastfeeding women
10. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving his consent
11. Known drug or alcohol abuse
12. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of study treatment (except local/topical or aerosol steroids)
13. Has a known history of active tuberculosis (Mycobacterium tuberculosis)
14. Has had a prior monoclonal antibody within 4 weeks or 5 half-life time (whichever is shorter) prior to the first dose of study treatment or who has not recovered (i.e., ≥ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
15. Has an active autoimmune / immune mediated inflammatory disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjörgen's syndrome will not be excluded from the study.
16. Has evidence of interstitial lung disease or active, non-infectious pneumonitis
17. Has an active infection requiring systemic therapy
18. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
19. Positive for Human Immunodeficiency Virus (HIV) antibody testing
20. Active or chronic hepatitis C and/or B infection. Patients with past/resolved HBV infection (defined as the presence of anti-hepatitis B core antibody, IgG anti-HBs +) are eligible. Hepatitis B virus DNA should be obtained in these patients prior to the first dose of study treatment. Patients positive for hepatitis C virus antibody are eligible only if PCR is negative for HCV RNA
21. Patients with altered hematopoietic or organ function, as indicated by the following criteria (assessed within 5 days prior registration):

    * White blood cell < 3000/μL
    * Polynuclear neutrophils < 1.5 x 109/L
    * Platelets < 100 x 109/L
    * Hemoglobin < 7.0 g/mL
    * Alanine aminotransferase/aspartate aminotransferase > 3.0 x ULN in the absence of liver metastases or > 5x upper limit of normal in the presence of liver metastases
    * Bilirubin > 1.5 x ULN (except Gilbert Syndrome: < 3.0 mg/dL)
    * Creatinine clearance ≤ 35 mL/min (measured or calculated by Cockcroft and Gault formula)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Objective response rate | at 8 weeks after diet initiation.
  Preliminary activity will be assessed by measuring objective response rate (ORR) (partial/complete response) of Nivolumab plus Ipilimumab concomitant to a special diet (KD continuous or discontinuous) or standard diet (SD) with or without (BHB) according to RECIST v1.1 at 8 weeks.

SECONDARY OUTCOMES:
Safety of Nivolumab plus Ipilimumab concomitant to a special diet | Events reported from the first day of diet and up to and including 100 days following the last day of diet could be included in estimating this incidence rate.
  the safety of Nivolumab plus Ipilimumab concomitant to a special diet (ketogenic diet, continuous or discontinuous) or standard diet (SD) with or without BHB will be measured by the rate of all and grade 3-4 adverse events (AEs) according to CTCAEv4, and compare the rate to historical data.
Assessment of weight | from the first day of diet and up to 2 years from diet initiation
  Assessment of weight in kilograms by baseline test and follow up in order to evaluate the impact of the diet concomitant to immunotherapy on nutritional status, muscle mass, and sarcopenia.
Assessment of albuminemia | from the first day of diet and up to 2 years from diet initiation
  Assessment of albuminemia in g/L in order to evaluate the impact of the diet concomitant to immunotherapy on nutritional status, muscle mass, and sarcopenia.
Assessment of prealbuminemia | from the first day of diet and up to 2 years from diet initiation
  Assessment of prealbuminemia in g/L in order to evaluate the impact of the diet concomitant to immunotherapy on nutritional status, muscle mass, and sarcopenia.
Assessment of C reactive protein | from the first day of diet and up to 2 years from diet initiation
  Assessment of C reactive protein in mg/L in order to evaluate the impact of the diet concomitant to immunotherapy on nutritional status, muscle mass, and sarcopenia.
Assessment of sarcopenia | from the first day of diet and up to 2 years from diet initiation
  Sarcopenia will be assessed according to SliceOmatic software V5.0 and preestablished thresholds of skeletal muscle tissue (-29 to +150 Hounsfield units). Axial L3 sections will be used to measure the total muscle area (TMA) and calculate skeletal muscle index (SMI, cm²/m²). Sarcopenia is defined as SMI lower than a sex-based threshold (<55.4 in men and <38.9 in women).
Assessment of Quality of Life (QoL) | At screening and 9 weeks after diet initiation
  explore the evolution of Patient Reported Outcomes using EORTC QLQ 30 file in all treated patients.
progression-free survival assessment | from the first day of diet and up to 2 years from diet initiation
  PFS is specified as the time between the date of the starting of the diet and the first date of documented progression, based on assessments (as per RECIST v1.1 criteria), or death due to any cause.
Sarcopenic event-free survival (SFS) | from the first day of diet and up to 2 years from diet initiation
  SFS will be estimated from intervention starting.
Overall survival (OS) | from the first day of diet and up to 2 years from diet initiation
  OS is specified as the time between the date of the starting of the diet and the date of the death whatever the cause.

CONTACTS AND LOCATIONS:
Overall Officials: Emeline COLOMBA BLAMEBLE, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (3):
- France (3):
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpitaux Cochin-Port-Royal, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dashti HM, Mathew TC, Hussein T, Asfar SK, Behbahani A, Khoursheed MA, Al-Sayer HM, Bo-Abbas YY, Al-Zaid NS. Long-term effects of a ketogenic diet in obese patients. Exp Clin Cardiol. 2004 Fall;9(3):200-5. PMID 19641727
- [Background] Woolf EC, Scheck AC. The ketogenic diet for the treatment of malignant glioma. J Lipid Res. 2015 Jan;56(1):5-10. doi: 10.1194/jlr.R046797. Epub 2014 Feb 6. PMID 24503133
- [Background] Chung HY, Park YK. Rationale, Feasibility and Acceptability of Ketogenic Diet for Cancer Treatment. J Cancer Prev. 2017 Sep;22(3):127-134. doi: 10.15430/JCP.2017.22.3.127. Epub 2017 Sep 30. PMID 29018777
- [Background] Levesque S, Pol JG, Ferrere G, Galluzzi L, Zitvogel L, Kroemer G. Trial watch: dietary interventions for cancer therapy. Oncoimmunology. 2019 Apr 3;8(7):1591878. doi: 10.1080/2162402X.2019.1591878. eCollection 2019. PMID 31143510
- [Background] Ferrere G, Tidjani Alou M, Liu P, Goubet AG, Fidelle M, Kepp O, Durand S, Iebba V, Fluckiger A, Daillere R, Thelemaque C, Grajeda-Iglesias C, Alves Costa Silva C, Aprahamian F, Lefevre D, Zhao L, Ryffel B, Colomba E, Arnedos M, Drubay D, Rauber C, Raoult D, Asnicar F, Spector T, Segata N, Derosa L, Kroemer G, Zitvogel L. Ketogenic diet and ketone bodies enhance the anticancer effects of PD-1 blockade. JCI Insight. 2021 Jan 25;6(2):e145207. doi: 10.1172/jci.insight.145207. PMID 33320838
- [Background] Motzer RJ, Tannir NM, McDermott DF, Aren Frontera O, Melichar B, Choueiri TK, Plimack ER, Barthelemy P, Porta C, George S, Powles T, Donskov F, Neiman V, Kollmannsberger CK, Salman P, Gurney H, Hawkins R, Ravaud A, Grimm MO, Bracarda S, Barrios CH, Tomita Y, Castellano D, Rini BI, Chen AC, Mekan S, McHenry MB, Wind-Rotolo M, Doan J, Sharma P, Hammers HJ, Escudier B; CheckMate 214 Investigators. Nivolumab plus Ipilimumab versus Sunitinib in Advanced Renal-Cell Carcinoma. N Engl J Med. 2018 Apr 5;378(14):1277-1290. doi: 10.1056/NEJMoa1712126. Epub 2018 Mar 21. PMID 29562145
- [Background] Motzer RJ, Rini BI, McDermott DF, Aren Frontera O, Hammers HJ, Carducci MA, Salman P, Escudier B, Beuselinck B, Amin A, Porta C, George S, Neiman V, Bracarda S, Tykodi SS, Barthelemy P, Leibowitz-Amit R, Plimack ER, Oosting SF, Redman B, Melichar B, Powles T, Nathan P, Oudard S, Pook D, Choueiri TK, Donskov F, Grimm MO, Gurney H, Heng DYC, Kollmannsberger CK, Harrison MR, Tomita Y, Duran I, Grunwald V, McHenry MB, Mekan S, Tannir NM; CheckMate 214 investigators. Nivolumab plus ipilimumab versus sunitinib in first-line treatment for advanced renal cell carcinoma: extended follow-up of efficacy and safety results from a randomised, controlled, phase 3 trial. Lancet Oncol. 2019 Oct;20(10):1370-1385. doi: 10.1016/S1470-2045(19)30413-9. Epub 2019 Aug 16. PMID 31427204
- [Background] Gianchecchi E, Fierabracci A. Inhibitory Receptors and Pathways of Lymphocytes: The Role of PD-1 in Treg Development and Their Involvement in Autoimmunity Onset and Cancer Progression. Front Immunol. 2018 Oct 17;9:2374. doi: 10.3389/fimmu.2018.02374. eCollection 2018. PMID 30386337
- [Background] Riley JL. PD-1 signaling in primary T cells. Immunol Rev. 2009 May;229(1):114-25. doi: 10.1111/j.1600-065X.2009.00767.x. PMID 19426218
- [Background] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Background] Lazar-Molnar E, Scandiuzzi L, Basu I, Quinn T, Sylvestre E, Palmieri E, Ramagopal UA, Nathenson SG, Guha C, Almo SC. Structure-guided development of a high-affinity human Programmed Cell Death-1: Implications for tumor immunotherapy. EBioMedicine. 2017 Mar;17:30-44. doi: 10.1016/j.ebiom.2017.02.004. Epub 2017 Feb 6. PMID 28233730
- [Background] Doherty JR, Cleveland JL. Targeting lactate metabolism for cancer therapeutics. J Clin Invest. 2013 Sep;123(9):3685-92. doi: 10.1172/JCI69741. Epub 2013 Sep 3. PMID 23999443
- [Background] Allen BG, Bhatia SK, Anderson CM, Eichenberger-Gilmore JM, Sibenaller ZA, Mapuskar KA, Schoenfeld JD, Buatti JM, Spitz DR, Fath MA. Ketogenic diets as an adjuvant cancer therapy: History and potential mechanism. Redox Biol. 2014;2:963-70. doi: 10.1016/j.redox.2014.08.002. Epub 2014 Aug 7. PMID 25460731
- [Background] Aykin-Burns N, Ahmad IM, Zhu Y, Oberley LW, Spitz DR. Increased levels of superoxide and H2O2 mediate the differential susceptibility of cancer cells versus normal cells to glucose deprivation. Biochem J. 2009 Feb 15;418(1):29-37. doi: 10.1042/BJ20081258. PMID 18937644
- [Background] Zhou Z, Hagopian K, Roberts M, et al. A Ketogenic Diet Increases Markers of Mitochondrial Content in a Tissue Specific Manner in Adult Mice. FASEB J. 2017;31(1_supplement):lb482-lb482. doi:10.1096/fasebj.31.1_supplement.lb482
- [Background] Stafford P, Abdelwahab MG, Kim DY, Preul MC, Rho JM, Scheck AC. The ketogenic diet reverses gene expression patterns and reduces reactive oxygen species levels when used as an adjuvant therapy for glioma. Nutr Metab (Lond). 2010 Sep 10;7:74. doi: 10.1186/1743-7075-7-74. PMID 20831808
- [Background] Cavaleri F, Bashar E. Potential Synergies of beta-Hydroxybutyrate and Butyrate on the Modulation of Metabolism, Inflammation, Cognition, and General Health. J Nutr Metab. 2018 Apr 1;2018:7195760. doi: 10.1155/2018/7195760. eCollection 2018. PMID 29805804
- [Background] Kimura I, Inoue D, Maeda T, Hara T, Ichimura A, Miyauchi S, Kobayashi M, Hirasawa A, Tsujimoto G. Short-chain fatty acids and ketones directly regulate sympathetic nervous system via G protein-coupled receptor 41 (GPR41). Proc Natl Acad Sci U S A. 2011 May 10;108(19):8030-5. doi: 10.1073/pnas.1016088108. Epub 2011 Apr 25. PMID 21518883
- [Background] Rahman M, Muhammad S, Khan MA, Chen H, Ridder DA, Muller-Fielitz H, Pokorna B, Vollbrandt T, Stolting I, Nadrowitz R, Okun JG, Offermanns S, Schwaninger M. The beta-hydroxybutyrate receptor HCA2 activates a neuroprotective subset of macrophages. Nat Commun. 2014 May 21;5:3944. doi: 10.1038/ncomms4944. PMID 24845831
- [Background] Youm YH, Nguyen KY, Grant RW, Goldberg EL, Bodogai M, Kim D, D'Agostino D, Planavsky N, Lupfer C, Kanneganti TD, Kang S, Horvath TL, Fahmy TM, Crawford PA, Biragyn A, Alnemri E, Dixit VD. The ketone metabolite beta-hydroxybutyrate blocks NLRP3 inflammasome-mediated inflammatory disease. Nat Med. 2015 Mar;21(3):263-9. doi: 10.1038/nm.3804. Epub 2015 Feb 16. PMID 25686106
- [Background] Shimazu T, Hirschey MD, Newman J, He W, Shirakawa K, Le Moan N, Grueter CA, Lim H, Saunders LR, Stevens RD, Newgard CB, Farese RV Jr, de Cabo R, Ulrich S, Akassoglou K, Verdin E. Suppression of oxidative stress by beta-hydroxybutyrate, an endogenous histone deacetylase inhibitor. Science. 2013 Jan 11;339(6116):211-4. doi: 10.1126/science.1227166. Epub 2012 Dec 6. PMID 23223453
- [Background] Xie G, Zhou Q, Qiu CZ, Dai WK, Wang HP, Li YH, Liao JX, Lu XG, Lin SF, Ye JH, Ma ZY, Wang WJ. Ketogenic diet poses a significant effect on imbalanced gut microbiota in infants with refractory epilepsy. World J Gastroenterol. 2017 Sep 7;23(33):6164-6171. doi: 10.3748/wjg.v23.i33.6164. PMID 28970732
- [Background] Braun S, Bitton-Worms K, LeRoith D. The link between the metabolic syndrome and cancer. Int J Biol Sci. 2011;7(7):1003-15. doi: 10.7150/ijbs.7.1003. Epub 2011 Aug 16. PMID 21912508
- [Background] Tracz AF, Szczylik C, Porta C, Czarnecka AM. Insulin-like growth factor-1 signaling in renal cell carcinoma. BMC Cancer. 2016 Jul 12;16:453. doi: 10.1186/s12885-016-2437-4. PMID 27405474
- [Background] Hakimi AA, Reznik E, Lee CH, Creighton CJ, Brannon AR, Luna A, Aksoy BA, Liu EM, Shen R, Lee W, Chen Y, Stirdivant SM, Russo P, Chen YB, Tickoo SK, Reuter VE, Cheng EH, Sander C, Hsieh JJ. An Integrated Metabolic Atlas of Clear Cell Renal Cell Carcinoma. Cancer Cell. 2016 Jan 11;29(1):104-116. doi: 10.1016/j.ccell.2015.12.004. PMID 26766592
- [Background] Zhang X, Tang N, Hadden TJ, Rishi AK. Akt, FoxO and regulation of apoptosis. Biochim Biophys Acta. 2011 Nov;1813(11):1978-86. doi: 10.1016/j.bbamcr.2011.03.010. Epub 2011 Mar 31. PMID 21440011
- [Background] Furusawa Y, Obata Y, Fukuda S, Endo TA, Nakato G, Takahashi D, Nakanishi Y, Uetake C, Kato K, Kato T, Takahashi M, Fukuda NN, Murakami S, Miyauchi E, Hino S, Atarashi K, Onawa S, Fujimura Y, Lockett T, Clarke JM, Topping DL, Tomita M, Hori S, Ohara O, Morita T, Koseki H, Kikuchi J, Honda K, Hase K, Ohno H. Commensal microbe-derived butyrate induces the differentiation of colonic regulatory T cells. Nature. 2013 Dec 19;504(7480):446-50. doi: 10.1038/nature12721. Epub 2013 Nov 13. PMID 24226770
- [Background] O'Flanagan CH, Smith LA, McDonell SB, Hursting SD. When less may be more: calorie restriction and response to cancer therapy. BMC Med. 2017 May 24;15(1):106. doi: 10.1186/s12916-017-0873-x. PMID 28539118
- [Background] Baranano KW, Hartman AL. The ketogenic diet: uses in epilepsy and other neurologic illnesses. Curr Treat Options Neurol. 2008 Nov;10(6):410-9. doi: 10.1007/s11940-008-0043-8. PMID 18990309
- [Background] Noakes TD. Low-carbohydrate and high-fat intake can manage obesity and associated conditions: occasional survey. S Afr Med J. 2013 Sep 30;103(11):826-30. doi: 10.7196/samj.7302. PMID 24148165
- [Background] McNally MA, Hartman AL. Ketone bodies in epilepsy. J Neurochem. 2012 Apr;121(1):28-35. doi: 10.1111/j.1471-4159.2012.07670.x. Epub 2012 Feb 7. PMID 22268909
- [Background] Cox PJ, Kirk T, Ashmore T, Willerton K, Evans R, Smith A, Murray AJ, Stubbs B, West J, McLure SW, King MT, Dodd MS, Holloway C, Neubauer S, Drawer S, Veech RL, Griffin JL, Clarke K. Nutritional Ketosis Alters Fuel Preference and Thereby Endurance Performance in Athletes. Cell Metab. 2016 Aug 9;24(2):256-68. doi: 10.1016/j.cmet.2016.07.010. Epub 2016 Jul 27. PMID 27475046
- [Background] Lambrechts DA, Bovens MJ, de la Parra NM, Hendriksen JG, Aldenkamp AP, Majoie MJ. Ketogenic diet effects on cognition, mood, and psychosocial adjustment in children. Acta Neurol Scand. 2013 Feb;127(2):103-8. doi: 10.1111/j.1600-0404.2012.01686.x. Epub 2012 Jun 12. PMID 22690843
- [Background] Newport MT, VanItallie TB, Kashiwaya Y, King MT, Veech RL. A new way to produce hyperketonemia: use of ketone ester in a case of Alzheimer's disease. Alzheimers Dement. 2015 Jan;11(1):99-103. doi: 10.1016/j.jalz.2014.01.006. Epub 2014 Oct 7. PMID 25301680
- [Background] Westman EC, Feinman RD, Mavropoulos JC, Vernon MC, Volek JS, Wortman JA, Yancy WS, Phinney SD. Low-carbohydrate nutrition and metabolism. Am J Clin Nutr. 2007 Aug;86(2):276-84. doi: 10.1093/ajcn/86.2.276. PMID 17684196
- [Background] Paoli A, Rubini A, Volek JS, Grimaldi KA. Beyond weight loss: a review of the therapeutic uses of very-low-carbohydrate (ketogenic) diets. Eur J Clin Nutr. 2013 Aug;67(8):789-96. doi: 10.1038/ejcn.2013.116. Epub 2013 Jun 26. PMID 23801097
- [Background] Schmidt M, Pfetzer N, Schwab M, Strauss I, Kammerer U. Effects of a ketogenic diet on the quality of life in 16 patients with advanced cancer: A pilot trial. Nutr Metab (Lond). 2011 Jul 27;8(1):54. doi: 10.1186/1743-7075-8-54. PMID 21794124
- [Background] Soto-Mota A, Vansant H, Evans RD, Clarke K. Safety and tolerability of sustained exogenous ketosis using ketone monoester drinks for 28 days in healthy adults. Regul Toxicol Pharmacol. 2019 Dec;109:104506. doi: 10.1016/j.yrtph.2019.104506. Epub 2019 Oct 23. PMID 31655093
- [Background] Klement RJ, Champ CE, Otto C, Kammerer U. Anti-Tumor Effects of Ketogenic Diets in Mice: A Meta-Analysis. PLoS One. 2016 May 9;11(5):e0155050. doi: 10.1371/journal.pone.0155050. eCollection 2016. PMID 27159218
- [Background] Maurer GD, Brucker DP, Bahr O, Harter PN, Hattingen E, Walenta S, Mueller-Klieser W, Steinbach JP, Rieger J. Differential utilization of ketone bodies by neurons and glioma cell lines: a rationale for ketogenic diet as experimental glioma therapy. BMC Cancer. 2011 Jul 26;11:315. doi: 10.1186/1471-2407-11-315. PMID 21791085
- [Background] Seyfried TN, Sanderson TM, El-Abbadi MM, McGowan R, Mukherjee P. Role of glucose and ketone bodies in the metabolic control of experimental brain cancer. Br J Cancer. 2003 Oct 6;89(7):1375-82. doi: 10.1038/sj.bjc.6601269. PMID 14520474
- [Background] Otto C, Kaemmerer U, Illert B, Muehling B, Pfetzer N, Wittig R, Voelker HU, Thiede A, Coy JF. Growth of human gastric cancer cells in nude mice is delayed by a ketogenic diet supplemented with omega-3 fatty acids and medium-chain triglycerides. BMC Cancer. 2008 Apr 30;8:122. doi: 10.1186/1471-2407-8-122. PMID 18447912
- [Background] Freedland SJ, Mavropoulos J, Wang A, Darshan M, Demark-Wahnefried W, Aronson WJ, Cohen P, Hwang D, Peterson B, Fields T, Pizzo SV, Isaacs WB. Carbohydrate restriction, prostate cancer growth, and the insulin-like growth factor axis. Prostate. 2008 Jan 1;68(1):11-9. doi: 10.1002/pros.20683. PMID 17999389
- [Background] Abdelwahab MG, Fenton KE, Preul MC, Rho JM, Lynch A, Stafford P, Scheck AC. The ketogenic diet is an effective adjuvant to radiation therapy for the treatment of malignant glioma. PLoS One. 2012;7(5):e36197. doi: 10.1371/journal.pone.0036197. Epub 2012 May 1. PMID 22563484
- [Background] Zahra A, Fath MA, Opat E, Mapuskar KA, Bhatia SK, Ma DC, Rodman SN III, Snyders TP, Chenard CA, Eichenberger-Gilmore JM, Bodeker KL, Ahmann L, Smith BJ, Vollstedt SA, Brown HA, Hejleh TA, Clamon GH, Berg DJ, Szweda LI, Spitz DR, Buatti JM, Allen BG. Consuming a Ketogenic Diet while Receiving Radiation and Chemotherapy for Locally Advanced Lung Cancer and Pancreatic Cancer: The University of Iowa Experience of Two Phase 1 Clinical Trials. Radiat Res. 2017 Jun;187(6):743-754. doi: 10.1667/RR14668.1. Epub 2017 Apr 24. PMID 28437190
- [Background] Galland L. The gut microbiome and the brain. J Med Food. 2014 Dec;17(12):1261-72. doi: 10.1089/jmf.2014.7000. PMID 25402818
- [Background] Vetizou M, Pitt JM, Daillere R, Lepage P, Waldschmitt N, Flament C, Rusakiewicz S, Routy B, Roberti MP, Duong CP, Poirier-Colame V, Roux A, Becharef S, Formenti S, Golden E, Cording S, Eberl G, Schlitzer A, Ginhoux F, Mani S, Yamazaki T, Jacquelot N, Enot DP, Berard M, Nigou J, Opolon P, Eggermont A, Woerther PL, Chachaty E, Chaput N, Robert C, Mateus C, Kroemer G, Raoult D, Boneca IG, Carbonnel F, Chamaillard M, Zitvogel L. Anticancer immunotherapy by CTLA-4 blockade relies on the gut microbiota. Science. 2015 Nov 27;350(6264):1079-84. doi: 10.1126/science.aad1329. Epub 2015 Nov 5. PMID 26541610
- [Background] Routy B, Le Chatelier E, Derosa L, Duong CPM, Alou MT, Daillere R, Fluckiger A, Messaoudene M, Rauber C, Roberti MP, Fidelle M, Flament C, Poirier-Colame V, Opolon P, Klein C, Iribarren K, Mondragon L, Jacquelot N, Qu B, Ferrere G, Clemenson C, Mezquita L, Masip JR, Naltet C, Brosseau S, Kaderbhai C, Richard C, Rizvi H, Levenez F, Galleron N, Quinquis B, Pons N, Ryffel B, Minard-Colin V, Gonin P, Soria JC, Deutsch E, Loriot Y, Ghiringhelli F, Zalcman G, Goldwasser F, Escudier B, Hellmann MD, Eggermont A, Raoult D, Albiges L, Kroemer G, Zitvogel L. Gut microbiome influences efficacy of PD-1-based immunotherapy against epithelial tumors. Science. 2018 Jan 5;359(6371):91-97. doi: 10.1126/science.aan3706. Epub 2017 Nov 2. PMID 29097494
- [Background] Gopalakrishnan V, Spencer CN, Nezi L, Reuben A, Andrews MC, Karpinets TV, Prieto PA, Vicente D, Hoffman K, Wei SC, Cogdill AP, Zhao L, Hudgens CW, Hutchinson DS, Manzo T, Petaccia de Macedo M, Cotechini T, Kumar T, Chen WS, Reddy SM, Szczepaniak Sloane R, Galloway-Pena J, Jiang H, Chen PL, Shpall EJ, Rezvani K, Alousi AM, Chemaly RF, Shelburne S, Vence LM, Okhuysen PC, Jensen VB, Swennes AG, McAllister F, Marcelo Riquelme Sanchez E, Zhang Y, Le Chatelier E, Zitvogel L, Pons N, Austin-Breneman JL, Haydu LE, Burton EM, Gardner JM, Sirmans E, Hu J, Lazar AJ, Tsujikawa T, Diab A, Tawbi H, Glitza IC, Hwu WJ, Patel SP, Woodman SE, Amaria RN, Davies MA, Gershenwald JE, Hwu P, Lee JE, Zhang J, Coussens LM, Cooper ZA, Futreal PA, Daniel CR, Ajami NJ, Petrosino JF, Tetzlaff MT, Sharma P, Allison JP, Jenq RR, Wargo JA. Gut microbiome modulates response to anti-PD-1 immunotherapy in melanoma patients. Science. 2018 Jan 5;359(6371):97-103. doi: 10.1126/science.aan4236. Epub 2017 Nov 2. PMID 29097493
- [Background] Matson V, Fessler J, Bao R, Chongsuwat T, Zha Y, Alegre ML, Luke JJ, Gajewski TF. The commensal microbiome is associated with anti-PD-1 efficacy in metastatic melanoma patients. Science. 2018 Jan 5;359(6371):104-108. doi: 10.1126/science.aao3290. PMID 29302014
- [Background] Derosa L, Routy B, Fidelle M, Iebba V, Alla L, Pasolli E, Segata N, Desnoyer A, Pietrantonio F, Ferrere G, Fahrner JE, Le Chatellier E, Pons N, Galleron N, Roume H, Duong CPM, Mondragon L, Iribarren K, Bonvalet M, Terrisse S, Rauber C, Goubet AG, Daillere R, Lemaitre F, Reni A, Casu B, Alou MT, Alves Costa Silva C, Raoult D, Fizazi K, Escudier B, Kroemer G, Albiges L, Zitvogel L. Gut Bacteria Composition Drives Primary Resistance to Cancer Immunotherapy in Renal Cell Carcinoma Patients. Eur Urol. 2020 Aug;78(2):195-206. doi: 10.1016/j.eururo.2020.04.044. Epub 2020 May 4. PMID 32376136
- [Background] Salgia NJ, Bergerot PG, Maia MC, Dizman N, Hsu J, Gillece JD, Folkerts M, Reining L, Trent J, Highlander SK, Pal SK. Stool Microbiome Profiling of Patients with Metastatic Renal Cell Carcinoma Receiving Anti-PD-1 Immune Checkpoint Inhibitors. Eur Urol. 2020 Oct;78(4):498-502. doi: 10.1016/j.eururo.2020.07.011. Epub 2020 Aug 19. PMID 32828600
- [Background] Desilets A, Elkrief A, Routy B. The Link Between the Gut Microbiome and Response to Immune Checkpoint Inhibitors in Renal Cell Carcinoma. Eur Urol. 2021 Jan;79(1):1-2. doi: 10.1016/j.eururo.2020.09.001. Epub 2020 Sep 16. No abstract available. PMID 32950294
- [Background] Daillere R, Derosa L, Bonvalet M, Segata N, Routy B, Gariboldi M, Budinska E, De Vries IJM, Naccarati AG, Zitvogel V, Caldas C, Engstrand L, Loilbl S, Fieschi J, Heinzerling L, Kroemer G, Zitvogel L. Trial watch : the gut microbiota as a tool to boost the clinical efficacy of anticancer immunotherapy. Oncoimmunology. 2020 Jun 3;9(1):1774298. doi: 10.1080/2162402X.2020.1774298. PMID 32934879
- [Background] Liu H, Wang J, He T, Becker S, Zhang G, Li D, Ma X. Butyrate: A Double-Edged Sword for Health? Adv Nutr. 2018 Jan 1;9(1):21-29. doi: 10.1093/advances/nmx009. PMID 29438462
- [Background] Schwartz S, Friedberg I, Ivanov IV, Davidson LA, Goldsby JS, Dahl DB, Herman D, Wang M, Donovan SM, Chapkin RS. A metagenomic study of diet-dependent interaction between gut microbiota and host in infants reveals differences in immune response. Genome Biol. 2012 Apr 30;13(4):r32. doi: 10.1186/gb-2012-13-4-r32. PMID 22546241
- [Background] Swidsinski A, Dorffel Y, Loening-Baucke V, Gille C, Goktas O, Reisshauer A, Neuhaus J, Weylandt KH, Guschin A, Bock M. Reduced Mass and Diversity of the Colonic Microbiome in Patients with Multiple Sclerosis and Their Improvement with Ketogenic Diet. Front Microbiol. 2017 Jun 28;8:1141. doi: 10.3389/fmicb.2017.01141. eCollection 2017. PMID 28702003
- [Background] McGettrick AF, O'Neill LA. How metabolism generates signals during innate immunity and inflammation. J Biol Chem. 2013 Aug 9;288(32):22893-8. doi: 10.1074/jbc.R113.486464. Epub 2013 Jun 24. PMID 23798679
- [Background] Lussier DM, Woolf EC, Johnson JL, Brooks KS, Blattman JN, Scheck AC. Enhanced immunity in a mouse model of malignant glioma is mediated by a therapeutic ketogenic diet. BMC Cancer. 2016 May 13;16:310. doi: 10.1186/s12885-016-2337-7. PMID 27178315
- [Background] Hussain TA, Mathew TC, Dashti AA, Asfar S, Al-Zaid N, Dashti HM. Effect of low-calorie versus low-carbohydrate ketogenic diet in type 2 diabetes. Nutrition. 2012 Oct;28(10):1016-21. doi: 10.1016/j.nut.2012.01.016. Epub 2012 Jun 5. PMID 22673594
- [Background] Gubin MM, Zhang X, Schuster H, Caron E, Ward JP, Noguchi T, Ivanova Y, Hundal J, Arthur CD, Krebber WJ, Mulder GE, Toebes M, Vesely MD, Lam SS, Korman AJ, Allison JP, Freeman GJ, Sharpe AH, Pearce EL, Schumacher TN, Aebersold R, Rammensee HG, Melief CJ, Mardis ER, Gillanders WE, Artyomov MN, Schreiber RD. Checkpoint blockade cancer immunotherapy targets tumour-specific mutant antigens. Nature. 2014 Nov 27;515(7528):577-81. doi: 10.1038/nature13988. PMID 25428507
- [Background] Sucker A, Zhao F, Pieper N, Heeke C, Maltaner R, Stadtler N, Real B, Bielefeld N, Howe S, Weide B, Gutzmer R, Utikal J, Loquai C, Gogas H, Klein-Hitpass L, Zeschnigk M, Westendorf AM, Trilling M, Horn S, Schilling B, Schadendorf D, Griewank KG, Paschen A. Acquired IFNgamma resistance impairs anti-tumor immunity and gives rise to T-cell-resistant melanoma lesions. Nat Commun. 2017 May 31;8:15440. doi: 10.1038/ncomms15440. PMID 28561041
- [Background] Arumugam M, Raes J, Pelletier E, Le Paslier D, Yamada T, Mende DR, Fernandes GR, Tap J, Bruls T, Batto JM, Bertalan M, Borruel N, Casellas F, Fernandez L, Gautier L, Hansen T, Hattori M, Hayashi T, Kleerebezem M, Kurokawa K, Leclerc M, Levenez F, Manichanh C, Nielsen HB, Nielsen T, Pons N, Poulain J, Qin J, Sicheritz-Ponten T, Tims S, Torrents D, Ugarte E, Zoetendal EG, Wang J, Guarner F, Pedersen O, de Vos WM, Brunak S, Dore J; MetaHIT Consortium; Antolin M, Artiguenave F, Blottiere HM, Almeida M, Brechot C, Cara C, Chervaux C, Cultrone A, Delorme C, Denariaz G, Dervyn R, Foerstner KU, Friss C, van de Guchte M, Guedon E, Haimet F, Huber W, van Hylckama-Vlieg J, Jamet A, Juste C, Kaci G, Knol J, Lakhdari O, Layec S, Le Roux K, Maguin E, Merieux A, Melo Minardi R, M'rini C, Muller J, Oozeer R, Parkhill J, Renault P, Rescigno M, Sanchez N, Sunagawa S, Torrejon A, Turner K, Vandemeulebrouck G, Varela E, Winogradsky Y, Zeller G, Weissenbach J, Ehrlich SD, Bork P. Enterotypes of the human gut microbiome. Nature. 2011 May 12;473(7346):174-80. doi: 10.1038/nature09944. Epub 2011 Apr 20. PMID 21508958
- [Background] Belizario JE, Napolitano M. Human microbiomes and their roles in dysbiosis, common diseases, and novel therapeutic approaches. Front Microbiol. 2015 Oct 6;6:1050. doi: 10.3389/fmicb.2015.01050. eCollection 2015. PMID 26500616